CLINICAL TRIAL: NCT04545879
Title: Investigating the Gut Microbiota Modulation Effects of Allicin for Cardiovascular Disease Protection and Establishing Microbiota Directed Personalized Nutrition Guidance With Novel Humanized Gnotobiotic Mice Model, Microbial Culturomics and Metabolomic Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 201712031RIND
Record Dates: First submitted 2020-09-06; First posted 2020-09-11 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2019-02

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Raw garlic juice (Experimental): Raw garlic juice treatment group
  Interventions: Dietary Supplement: Raw garlic juice containing allicin

INTERVENTIONS:
Dietary Supplement: Raw garlic juice containing allicin — Fresh garlic juice containing around 48mg allicin for 7 days

SUMMARY:
Investigators recruited 10 trimethylamine N-oxide (TMAO) producers to test the effect of garlic juice containing allicin on gut microbiota modulation and TMAO production.

DETAILED DESCRIPTION:
Trimethylamine N-oxide (TMAO) was recently discovered as a novel and independent risk factor for promoting atherosclerosis while it is generated from dietary carnitine through the metabolism of gut microbiota for decades. Allicin, the major compound in raw garlic juice, is a naturally antimicrobial phytochemical found in raw garlic juice and easily acquired from the diet. Investigators' previous study suggests dietary allicin reduces the transformation of L-carnitine to TMAO through the impact on gut microbiota in mice. Therefore, it is worth investigating whether raw garlic juice intake could reduce the TMAO productivity of human gut microbiota as well as modulate gut microflora. Investigators plan to recruit 10 TMAO producers to receive garlic juice for one week. The plasma and urine TMAO concentration will be measured by the LC-MS, and the gut microbiota composition will be analyzed by the next-generation sequencing, through bioinformatics analysis. Investigators expected after intake garlic juice for one week, it could prevent the cardiovascular disease risk via gut microbiota modulation and reduction of plasma and urine TMAO.

Screening of the TMAO producer:

The healthy participants were recruited, the criteria as follows: (1) age ≥ 20 years old; (2) no exposure to antibiotics, probiotics, or carnitine supplements within the previous month; (3) have no history of chronic diseases including, diabetes mellitus, myasthenia gravis, chronic renal disease, hyperparathyroidism, epilepsy, and severe anemia; (4) Participants were excluded from the study if they reported recent gastrointestinal discomfort (such as abdominal pain or diarrhea). To screening the TMAO producer, Investigators use the oral carnitine challenge test (OCCT) method which previously exhibited better efficacy than fasting plasma TMAO to identify the TMAO producer phenotype. All of the participants fasted at least 8 hours before performing OCCT. 1500 mg of L-carnitine (3 tablets, General Nutrition Centers, Inc., USA) orally administrated to the participants. The blood and urine of participants were collected at 0, 24, 48, and 72 hours after carnitine intake. Participants with plasma TMAO ≧ 10 μM after OCCT were defined as high TMAO producers and proceeded into the garlic juice intervention test.

Garlic Juice Intervention:

High-TMAO producers asked to consume 55 mL of raw garlic juice (48 mg of allicin equivalent) once a day during dinner for one week. High-TMAO producers suggested consuming the garlic juice with a meal. The high-TMAO producers were free to choose their diet, no restriction on the type of food. After one week of raw garlic juice intervention, the second OCCT was performed.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-65 years old
* Healthy subjects with TMAO producing ability

Exclusion Criteria:

* Exposure to antibiotics, probiotics, or carnitine supplements within the previous month
* Have a history of chronic diseases including, diabetes mellitus, myasthenia gravis, chronic renal disease, hyperparathyroidism, epilepsy, and severe anemia
* Have gastrointestinal discomfort (such as abdominal pain or diarrhea)

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2019-05-18 (Actual); Study Completion 2019-05-18 (Actual)

PRIMARY OUTCOMES:
Plasma and urine TMAO level (ppm) | 6 months
  Quantitation of plasma and urine TMAO level by LC-MS
Compositional analysis of gut microbiota (% of different bacteria species) | 6 months
  Next-generation sequencing and bioinformatics

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Shiang Wu, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan